CLINICAL TRIAL: NCT00044382
Title: A Phase II Open Label Study of the Safety and Efficacy of CC-5013 Treatment For Patients With Myelodysplastic Syndrome
Brief Title: Study of the Safety and Efficacy of CC-5013 Treatment For Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MDS-501-001
Record Dates: First submitted 2002-08-27; First posted 2002-08-29 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndrome
Keywords: Revimid; CC5013; CC-5013
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CC-5013

SUMMARY:
To estimate the percent of patients with myelodysplastic syndromes (MDS) who experience erythroid response and the interval to response with daily treatment of 25 mg of CC-5013 .

ELIGIBILITY:
* Diagnosis of de novo myelodysplastic syndrome of at least 12 weeks duration.
* Baseline mean hemoglobin < 10.0 g/dL (untransfused) and/or be transfusion dependent defined by requiring at least 4 units of RBC in the 8 weeks prior to baseline.
* More than 30 days must have elapsed since any previous treatment for MDS, other than transfusion.
* Women must not be pregnant or lactating
* No use of another experimental study drug within 30 dy\ays of baseline
* Understand and sign written informed consent
* Able to adhere to study visit schedule, understand and comply with other protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2002-02-01 (Actual); Primary Completion 2007-01-01 (Actual); Study Completion 2007-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Cancer Center, Tucson, Arizona, United States

REFERENCES:
- [Background] List A, Kurtin S, Roe DJ, Buresh A, Mahadevan D, Fuchs D, Rimsza L, Heaton R, Knight R, Zeldis JB. Efficacy of lenalidomide in myelodysplastic syndromes. N Engl J Med. 2005 Feb 10;352(6):549-57. doi: 10.1056/NEJMoa041668. PMID 15703420